CLINICAL TRIAL: NCT06204042
Title: Glanzmann Thrombasthenia Natural History Study+
Brief Title: Multinational Glanzmann Study
Acronym: Glanzmann-NHS
Status: Not yet recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Roger Schutgens, Prof. Dr. R.E.G. Schutgens, UMC Utrecht
Other Study IDs: NL85068.041.24
Record Dates: First submitted 2023-12-05; First posted 2024-01-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Glanzmann Thrombasthenia
MeSH Terms: conditions — Thrombasthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glanzmann thrombasthenia is a rare autosomal recessive platelet disorder characterized by a lack of functional integrins alfaIIb or beta3 (glycoproteins IIb/IIIa). The prevalence is variously reported to be between 1:200,000 to 1:1,000,000, with substantial geographic variation. The clinical phenotype is dominated by an increased mucocutaneous bleeding tendency. In absence of a primary bleeding prophylaxis, the current treatment of Glanzmann thrombasthenia is mainly focused on prevention or management of bleeding. However, as potential new therapies emerge, clinicians require unbiased, long-term safety and efficacy data for both current treatment and new therapies.

We have designed this study to investigate genetic phenotype (ITGA2B and ITGB3 genes) and the prevalence of antibodies against human leucocyte antigen (HLA) and human platelet antigen (HPA), the latter two being a potential consequence of the current golden standard treatment: platelet transfusion. The results of this study will be merged with a longitudinal registry with retrospective and prospective data collection of clinical phenotype, haemorrhagic burden and bleeding management. Analysis of the data from the Glanzmann-NHS+ study and the registry will help us to get a better understanding of the clinical variation among participants with Glanzmann thrombasthenia. The ultimate goal is to accelerate improvement in the care of patients with Glanzmann thrombasthenia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥16 years);
* Biochemically or genetically diagnosed Glanzmann thrombasthenia.
* Willing and able to give written informed consent.

Exclusion Criteria:

* Patients with acquired thrombasthenic states caused by auto-immune disorders or drugs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with biochemically or genetically diagnosed Glanzmann thrombasthenia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Genetic analysis for Glanzmann thrombasthenia | Single measurement at Baseline
  Description of mutation analysis in the ITGA2B and ITGB3 genes.

SECONDARY OUTCOMES:
Incidence of anti-Human Leucocyte Antigen (HLA) antibodies | Single measurement at Baseline
  Cross-sectional evaluation of existing antibodies against Human Leucocyte Antigen (HLA) type I.
Incidence of anti-Human Platelet Antigen (HPA) antibodies | Single measurement at Baseline
  Cross-sectional evaluation of existing antibodies against Human Platelet Antigen (HPA)